CLINICAL TRIAL: NCT02196376
Title: Assessment of Antibodies and Inflammatory Markers in Postural Tachycardia Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Satish R. Raj, Adjunct Associate Professor of Medicine and Pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 140671
Record Dates: First submitted 2014-07-15; First posted 2014-07-22 (Estimated); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
Keywords: Postural orthostatic syndrome; orthostatic intolerance; autonomic dysfunction
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance; Primary Dysautonomias | interventions — Health Records, Personal; Restraint, Physical; Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood will be drawn for future assay and analysis of the following tests:
  Antibodies regulating cardiovascular function
  The clinical significance of these antibodies is unknown. We will share the results of the antibody panel with the subject, but with the caveat that no clinical interpretation or comment on significance can be made.
  Inflammatory markers
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- orthostatic tachycardia syndrome: participants with postural orthostatic tachycardia syndrome
  Interventions: Other: History; Other: Physical; Other: blood draw; Behavioral: Questionnaires
- control subjects: participants not diagnosed with postural orthostatic tachycardia syndrome
  Interventions: Other: History; Other: Physical; Other: blood draw; Behavioral: Questionnaires

INTERVENTIONS:
Other: History — the physician / PI will conduct a history that may include: demographics Framingham risk factors metabolic diseases inflammatory diseases autoimmune disorders review of medications date of last menstrual period (females) family history of autonomic disorders Onset of postural orthostatic tachycardia syndrome
Other: Physical — the physical exam will include: height weight orthostatic vitals (heart rate and blood pressure), supine and standing for up to 10 minutes.
  Beighton Criteria for Join Hypermobility Syndrome Dependent acrocyanosis
Other: blood draw — blood will be drawn for: antibodies regulating cardiovascular function inflammatory markers
  no more than 15 ml (1 TBSP) will be drawn.
Behavioral: Questionnaires — The questionnaires will be completed directly online (web-based interface) using a personalized link that will be provided to the subjects after they give their informed consent. These will be created in a REDCap-Survey environment, with the data collected and stored on a password-protected, HIPAA-compliant, secure computer server.
  The following questionnaires will be conducted:
  RAND-36 Health Thermometer Chalder Fatigue Scale Daily diary of Fatigue Symptoms - Fibromyalgia Pain Detect Questionnaire Orthostatic Grading Scale COMPASS-31

SUMMARY:
In this pilot study, the investigators will test the hypothesis that patients with postural tachycardia syndrome will have an elevated percentage of functional antibodies to adrenergic receptors compared with control subjects without POTS. The investigators further hypothesize that the percentage of POTS patients with antibodies will be higher in those patients with a viral infection at the onset of their illness than in those patients with other or undefined illness onsets.

DETAILED DESCRIPTION:
Postural orthostatic tachycardia syndrome is poorly understood. Many of these patients have elevated levels of plasma norepinephrine, particularly when upright One subgroup of patients has a primary hyperadrenergic state. The majority of patients have a marked deficit in plasma blood volume compared to healthy control subjects. The investigators have previously reported that some patients suffer paradoxically from a partial dysautonomia affecting the lower limbs. Most patients seem to suffer from either a primary or secondary increase in central sympathetic nervous system drive. Recent data have shown that patients with postural orthostatic tachycardia syndrome have a lower cardiac stroke volume than their healthy counterparts and this low stroke volume may drive their orthostatic tachycardia.

The investigators plan to do the following:

The physical examination will include (at minimum):

* Height
* Weight
* Orthostatic vital signs (heart rate and blood pressure) Supine and Standing for up to 10 minutes
* Beighton Criteria for Joint Hypermobility Syndrome (Ehlers-Danlos III)
* Dependent acrocyanosis (during stand test)

Continuous Heart Rate and Blood Pressure Recording A subset of subjects will be given the opportunity to also have continuous recordings of heart rate and blood pressure for 5-10 minutes while lying down quietly. They will be instrumented with EKG patches on their body and a finger blood pressure cuff, and these data will be digitally sampled and acquired on a dedicated laptop computer for later offline analysis.

There will be an optional rider on the consent form to allow the patient to consent to this portion of the study.

Blood work

Blood will be drawn for future assay and analysis of the following tests:

* Antibodies regulating cardiovascular function

  o The clinical significance of these antibodies is unknown. The investigators will share the results of the antibody panel with the subject, but with the caveat that no clinical interpretation or comment on significance can be made.
* Inflammatory markers

The total amount of blood drawn for this project will be less than 15 ml.

Questionnaires

* RAND-36
* Health Thermometer
* Chandler Fatigue Scale
* Daily diary of Fatigue Symptoms - Fibromyalgia
* Pain Detect Questionnaire
* Orthostatic Grading Scale
* COMPASS-31
* Structured History (including some of the elements from section 6.1)

These questionnaires will be completed directly online (web-based interface) using a personalized link that will be provided to the subjects after they give their informed consent. These will be created in a REDCap-Survey environment, with the data collected and stored on a password-protected, HIPAA-compliant, secure computer server.

ELIGIBILITY:
Inclusion Criteria:

* Postural Tachycardia Syndrome
* Previously diagnosed with POTS
* Control Subjects
* Not diagnosed with POTS
* Age between 13-80 years
* Male and female subjects are eligible.
* Able and willing to provide informed consent

Exclusion Criteria:

* Inability to give, or withdrawal of, informed consent
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol.

Ages: 13 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Chronic orthostatic intolerance, sometimes known as the postural tachycardia syndrome (POTS), is the most common disorder among patients seen at several centers specializing in diseases of the autonomic nervous system.
  excessive increase in heart rate [>30 min-1] on standing associated with orthostatic symptoms [including palpitation, chest pain syndrome, dyspnea on standing, mental clouding and difficulties with concentration], in the absence of orthostatic hypotension. Orthostatic tachycardia can produce substantial disability among otherwise healthy people. Patients typically feel tired and run down. Many also report a myriad of symptoms that are hard to categorize, often involving fatigue. We and others have reported that patients had a diminished quality of life.
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2014-07; Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Ab titer in POTS patients compared to control subjects | One time only, at first visit
  The primary outcome measure will be the proportion of subjects with alpha-1 Ab titer. The primary comparison will be the proportion of Ab titers between POTS patients compared to control subjects.

SECONDARY OUTCOMES:
comparison of the number of POTS patients with viral based Ab versus non-viral based Ab | One time only - at first study visit
  Blood samples will be collected at study visit.
comparison of the number of POTS patients with and without Ehlers Danlos syndrome III | One time only - at first study visit
  Ehlers Danlos Syndrome will be assessed during the physical exam. The hypermobility assessment (Beighton Score) will be used.
comparison of the number of POTS patients with a history of autoimmune disorders versus no history of auto-immune disorders | One time only - at first study visit
  History of auto-immune disorders will be collected during the history and physical performed by the physician.
comparison of the number of POTS patients with fatigue versus no history of fatigue based on severity of impact on normal daily activities. | One time only - at first study visit
  Fatigue will be assessed using the RAND-36 Health Thermometer Chalder Scale of Fatigue, and Daily Diary of Fatigue.
comparison of pain in POTS patients versus non-POTS patients | One time only - at first study visit
  Pain will be assessed using Fibromyalgia Pain Detect Questionnaire, Orthostatic Grading Scale and COMPASS-31.

CONTACTS AND LOCATIONS:
Overall Officials: Satish Raj, MD, MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States